CLINICAL TRIAL: NCT02141880
Title: The Tailgate Study: A Pilot Study Measuring the Impact of Acute Alcohol Intake on Intrahepatic Lipid
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Elizabeth Parks, Professor, Nutrition & Exercise Physiology-MED, University of Missouri-Columbia
Other Study IDs: 1211233
Record Dates: First submitted 2014-05-14; First posted 2014-05-20 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment: All subjects will be under the same protocol which is eating and drinking on one afternoon.

SUMMARY:
College drinking associated with sporting events is characterized by excess alcohol, along with food intake, over the duration of hours has the potential to cause a build up of fat in the liver. Fatty liver can increase blood glucose concentrations leading to a prediabetes like state.

The present study will determine how overweight men respond to the over-consumption of alcohol/food to identify which characteristics might protect some men from fatty liver, while others might be more susceptible to this condition.

The goal of this work is to determine the direct impact of alcohol/food intake to cause acute fatty liver through the stimulation of de novo lipogenesis in 20 overweight, healthy men. Understanding individual susceptibility to alcohol-induced fatty liver will aid in the development of strategies designed to help people mitigate these risks.

Hypothesis is that 5h excess consumption of alcohol and food will increase liver triglycerides by 4% or more, in comparison to fasting state.

DETAILED DESCRIPTION:
Subjects will participate in a single screening visit and a 24 hours in-patient stay at the clinical research center for treatment and tests.

No drugs will be used in this study, however, amounts of alcohol will be consumed to achieve, and maintain a breath alcohol at the legal limit (0.10).

The goals are to quantitate the increase in lipogenesis due to acute alcohol/food intake and to determine the effects of acute alcohol/food intake on liver-triglycerides.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Age 21-40
* BMI 25.1-35.0 kg/m2
* Waste girth < 55 inches
* Nonsmoking
* Moderate consumer of alcohol
* Fasting blood glucose < 125 mg/dL, alanine transaminase activity < 40 milliunits/L, plasma triglycerides < 200 mg/dL
* Sedentary
* Free of metabolic disorders

Exclusion Criteria:

* BMI < 25.1 or > 35.0 kg/m2
* Waste girth of greater 55 inches
* Use of any tabacco product
* Fasting plasma glucose ≥125 mg/dL, alanine transaminase activity ≥ 40 milliunits/L, plasma triglycerides ≥125 mg/dL
* Physically active
* Diabetes or other diseases that impact blood glucose or lipids
* Fatty liver disease

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy and overweight sedentary men.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Liver triglycerides | will be measured before (fasting) and after 5 hours of alcohol consumption
  Liver fat will be measured twice in each subject via magnetic resonance spectroscopy, blood will be drawn hourly and metabolites will be measured enzymatically.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Parks, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No